CLINICAL TRIAL: NCT01095809
Title: Open , Randomized Study About Efficacy, Safety and Tolerability od Repeated Dosis of Intravitreous Bevacizumab in Patients With Uveitic Macular Oedema
Brief Title: Efficacy, Safety and Tolerability of Repeated Dosis of Intravitreous Bevacizumab in Uveitic Macular Oedema
Acronym: EBEV
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: New intraocular steroid in the market. Recruitment no longer ethical.
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Alfredo Manuel Adan Civera, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EBEV
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2010-12

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis | interventions — Bevacizumab; Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- bevacizumab (Experimental): intravitreous bevacizumab 2,5 mg at baseline, week 4 and 8. reinjection is required.
  Interventions: Drug: bevacizumab
- triamcinolone acetonide (Experimental): intravitreous triamcinolone 2 mg, frequency: 3 months
  Interventions: Drug: triamcinolone acetonide

INTERVENTIONS:
Drug: bevacizumab — 2.5mg at baseline, week 4 and 8. Beyond this initial period if needed reinjection criteria are described in protocol
  Arms: bevacizumab
Drug: triamcinolone acetonide — 2 mg at baseline; frequency every three months if needed. reinjection criteria are described in protocol
  Arms: triamcinolone acetonide

SUMMARY:
The purpose of this study is to determine whether intravitreous bevacizumab or intravitreous triamcinolone acetonide are effective and safe in the treatment of uveitic macular oedema

ELIGIBILITY:
Inclusion Criteria:

* adult patients with uveitis or retinal vasculitis with unilateral or bilateral macular oedema
* with macular thickness > 250 micra using OCT
* visual acuity at least 20/200
* with stable treatment with oral prednisone at least during 3 months, either oral ciclosporin or other immunomodulator to treat intraocular inflammatory disease
* patient that can follow study's requirements
* patient who consents to participate

Exclusion Criteria:

* presence of corneal or crystalline opacity preventing observation of fundus of eye
* patients requiring ocular surgery in next 3 months
* one-eyed
* pregnancy and child breastfeeding
* previous history of glaucoma
* on treatment woth an experimental ocular drug
* previous thromboembolism or receiving oral anticoagulant treatment
* vitrectomy
* patients with proved tractional macular pathology associated to macular oedema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-04; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Macular Thickness Measurements Using Stratus Optical Coherence Tomography | 48 weeks

SECONDARY OUTCOMES:
visual acuity | 48 weeks
intraocular pressure | 48 weeks
opacity crystalline | 48 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital de Son Dureta, Palma de Mallorca, Spain/ Baleares
  - Hospital Santa creu i Sant Pau, Barcelona, Spain/ Catalonia
  - Instituto Vissum Alicante, Alicante, Spain/ Com. Valenciana
  - Hospital Vall d'Hebron, Barcelona, Spain/Catalonia
  - Hospital Clinic of Barcelona, Barcelona, Spain/Catalonia